CLINICAL TRIAL: NCT04458337
Title: SURgical Outcomes in COvid Patients - the SUROCO Multicenter Cohort Study
Brief Title: SURgical Outcomes in COvid Patients - the SUROCO Multicenter Cohort Study (COVID-19)
Acronym: SUROCO
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); St. Justine's Hospital (Other); Institut de Cardiologie de Montréal (Unknown); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); CHU de Quebec-Universite Laval (Other); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Sponsor
Other Study IDs: 19.386
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-09

CONDITIONS: Covid-19; SARS-CoV2; Surgery; Surgical Procedure; Complications, Late Effect of Complications; Postoperative Complications
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 patients undergoing a surgical procedure: The investigators propose to conduct a prospective observational cohort study on all patients suspected or confirmed being infected to SARS-CoV-2, or recovered from SARS-CoV-2, undergoing a surgery.

SUMMARY:
Overall mortality of COVID-19 is variable and has been reported to be between less than 1% and 7%. Many authors around the world also reported data on hospitalization rate, need for intensive care unit (ICU) care and need for mechanical ventilation in SARS-CoV-2 infected patients. To provide anesthetic and surgical care to SARS-CoV-2 infected patients, many health workers have to organize surgical platforms, personal protections and in-hospital trajectories to prevent dissemination and cross-contamination. However, no data has been published on the surgical need of these patients, their postoperative outcomes and the impact they may have on the operating room.

Postoperative outcomes in SARS-CoV-2 infected patients seem to be variable. Expected benefits from a surgical procedure may be different in this population if their postoperative mortality is higher than expected. The association between preoperative characteristics and postoperative outcomes in this population has to be better defined.

There is a need to better quantify these and better inform use of surgical resources during a pandemic. To address this knowledge gap, the investigators propose to conduct a multicenter observational cohort study in SARS-CoV-2 infected patients undergoing a surgical procedure, as well as in those who have recovered from COVID-19.

DETAILED DESCRIPTION:
METHODS Objectives

Primary: To describe postoperative outcomes in patients with COVID-19 undergoing a surgical procedure and measure the association between presence of symptoms and postoperative outcomes.

Secondary: To describe postoperative outcomes in patients undergoing a surgical procedure after they have healed from COVID-19 and measure the association between time from first positive test and postoperative outcomes.

Tertiary: To compare outcomes between symptomatic and asymptomatic COVID-19 patients undergoing a surgery with those who have healed from it.

Exposure variables:

For the primary objective, the exposure of interest will be the presence of symptoms at time of surgery. For the secondary objective, the exposure will be the length of time between first COVID-19 positive test and the date of surgery. For the tertiary objective, the status of the disease will be our exposure of interest.

Variable definitions:

All COVID-19 variables will be based on the first day of diagnosis (either clinical or by RT-PCR from either an oronasopharyngeal swab or an endotracheal specimen). The investigators will also capture asymptomatic SARS-CoV-2 carrier. Recovery at surgery will be defined as having two negative SARS-CoV-2 PCR tests between the last positive one and the surgery, or 1 negative test and a clinically significant period without symptoms between the last positive test and the negative one or no negative test but considered as recovered by the clinical team because of complete symptoms resolution.Criteria for "healed" status changed in November 2020 and were less restrictive (as detailed in table 1 of the protocol). No minimal or maximal delay will be applied between SARS-COV-2 infection and surgery for inclusion.

Surgical disease will be defined as the one reported by the surgeon. Surgeries will be further categorized into the following categories: neurosurgical (head, neck and spine), cardiac, thoracic, major vascular (intrathoracic and/or intra-abdominal), non-vascular abdominal (laparotomy or laparoscopy), urogenital (urology and/or gynecology), non-spine orthopedics, peripheral vascular, ENT and other. Any neurosurgical, cardiac, thoracic, major vascular or non-vascular abdominal surgery will be defined as a major surgery. The investigators will capture the surgical approach (minimally invasive or invasive) and the urgent nature of the procedure. Minimally invasive surgery will be defined as a one that does not need to open an anatomical cavity (laparoscopy, thoracoscopy, endoluminal). Urgency of surgery will be defined as one that needs to be done within 24 hours (emergent or urgent), or can wait for more than 24 hours (non-urgent).

The investigators will measure hospital survival. The investigators will also capture survival up to 30 days and 6 months using regular hospital follow-up. The investigators will use existing definitions for the postoperative pulmonary complications outcome. Non-pulmonary infectious complications will be defined as any infection that needed antibiotics for more than 72 hours. Acute kidney injury will be defined by the creatinine difference of the KDIGO-AKI criteria. Myocardial infraction and stroke will be defined as reported by treating physicians. Mechanical ventilation will be defined as any mechanical support (non-invasive or invasive). All 30-day outcomes will include any day with the outcome and the 30-day organ dysfunction free days will use existing definitions.

Sample size:

The investigators plan a convenient sample size depending on the number of patients and center included. Inclusion will start on the 13th of March 2020.

Analyses:

Primary objective The investigaors will first conduct descriptive analyses of baseline characteristics and outcomes of COVID-19 confirmed patients based on the presence of symptoms at the time of surgery (symptomatic versus asymptomatic). The investigators will report descriptively the following outcomes in both patients' population: proportion of patients with pulmonary complications, thromboembolic complications, non-pulmonary infectious complications, need for a new postoperative ICU admission, mean hospital length of stay, 30-day mechanical ventilation free-days and 30-day organ dysfunction free days. . To evaluate if presence of symptoms is associated with hospital survival in SARS-COV2 infected patients for the primary analysis, investigators will fit a multivariable Cox model that will include presence of symptoms, preoperative hospitalization, preoperative respiratory support need (invasive mechanical ventilation, oxygen therapy, no oxygen), urgency of surgery, importance of surgery (major versus minor) as independent variables and a frailty factor as a center random effect. If too few events our observed, investigators will limit covariables in their model.

Secondary objective The investigators will report descriptively patients who have recovered by categorizing them based on the time since first positive test (categorized as 0-4 weeks, 4-8 weeks and > 8 weeks). The investigators will report the same outcomes as previously mentioned. To analyze the effect of recovery time on postoperative survival, the investigators will fit a similar multivariable survival model . The investigators will include time since first positive COVID-19 test, preoperative hospitalization, preoperative respiratory support need (invasive mechanical ventilation, oxygen therapy, no oxygen), urgency of surgery, importance of surgery (major versus minor) as independent variables and a frailty factor as a center random effect. Investigators will explore non-linear relationship between time and the outcome.

Tertiary objective The investigators will report descriptively patients who have recovered and asymptomatic COVID-19 patients. To compare if those two groups of patients are different regarding hospital survival, the investigators will fit a multivariable survival model that will include status (recovered versus asymptomatic carrier), preoperative hospitalization, preoperative respiratory support need (invasive mechanical ventilation, oxygen therapy, no oxygen), urgency of surgery, importance of surgery (major versus minor) as independent variables and a frailty factor as a center random effect.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing a surgery with either a SARS-CoV-2 clinical suspicion based on reported symptoms during the pandemic (fever, myalgia, fatigue, cough, dyspnea, respiratory failure, diarrhea, vomiting, abdominal pain) or without any suggestive symptoms AND a SARS-CoV-2 confirmed infection with RT-PCR before surgery or within 72 hours after surgery. Patients who have recovered from SARS-CoV-2 infection will also be included. All patients up to 30th day of April 2021 will be included.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (children and adults) confirmed being infected to SARS-CoV-2 will be included, as well as patients who have recovered, undergoing a surgical procedure in designated Canadian Centers. The investigators will include all patients up to 30th day of April 2021.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Hospital survival | 30 days post-operation
  Survival was calculated from the date of participant randomization to the date of participant death due to any cause. If the participant was discharged from the hospital and not seen afterwards, the date of hospital discharge was entered as the last day seen alive.

SECONDARY OUTCOMES:
Occurrence of postoperative respiratory complications | 30 days post-operation
  The respiratory complications were recorded as diagnosed by medical personnel and/or medical imaging. The complications included atelectasis, pneumonia, acute respiratory distress syndrome (ARDS) and pulmonary aspiration.
Occurrence of postoperative non-pulmonary infectious complications | 30 days post-operation
  The infection site complications were recorded as diagnosed by medical personnel and/or medical imaging. The infectious site included surgical incision or puncture site, surgical abscess, anastomotic leak, central nervous system, urinary tract infection, osteomyelitis, positive blood culture, etc. A postoperative infection had to be accompanied by an antimicrobial therapy lasting longer than 72 hours. In the event a patient suffered from two infections in the same site, both dates were recorded.
Occurrence of acute kidney injury (AKI) | 30 days post-operation
  The grade of AKI was classified according to the KDIGO-AKI criteria using the highest reported creatinine or the need for new renal replacement therapy after surgery, including any mode of renal replacement therapy.
Occurrence of postoperative thromboembolic complications | 30 days post-operation
  The thromboembolic complications were recorded as diagnosed by medical personnel and/or medical imaging. These included myocardial infarction, stroke, pulmonary embolism and cardiac arrest. Myocardial infarction was defined as a physician's diagnosis of a MI, which includes ST Elevation Myocardial Ischemia (STEMI) or Non-ST Elevation Myocardial Ischemia (NSTEMI).
The need for a new postoperative ICU admission | 30 days post-operation
  The dates for all ICU admissions and dates of ICU discharge were recorded. If the patient was readmitted to ICU following his initial admission to ICU, the dates for admissions and discharges were recorded.
Hospital length of stay | An average of 7 days
  The number of days of hospital length of stay was calculated using the difference between the local date of discharge from the hospital and the date of hospital admission (day of surgery if ambulatory surgery). If the patient died during surgery or prior to hospital discharge, the patient's date of death was recorded as the date of discharge.
30-day mechanical ventilation free-days | 30 days post-operation
  The total number of days the patient was on invasive mechanical support was recorded. If mechanical ventilation was weaned and started again, the days when the patients were under mechanical ventilation were indicated. Non-invasive ventilation or high-flow nasal cannula (HFNC) were not included.
30-day organ dysfunction free days | 30 days post-operation
  The total number of days the patient was: on invasive mechanical ventilator, under vasopressor therapy for more than 2 hours up to 30 days after surgery and spent under renal replacement therapy was recorded.
Surgical reinterventions | 30 days post-operation
  Any surgical reintervention in the operating room either related or unrelated to the initial intervention was recorded.
Any ICU admission during the index hospital stay | 30 days post-operation
  The dates for all ICU admissions and dates of ICU discharge were recorded. If the patient was admitted to ICU just after the index surgery, the date of ICU admission and time at which it occurred were recorded.
30-day survival | 30 days post-operation
  Survival was calculated from the date of participant randomization to the date of participant death due to any cause, within 30 days after the surgery.
6-month survival | 6 months post-operation
  Survival was calculated from the date of participant randomization to the date of participant death due to any cause, within 6 months after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: François-Martin Carrier, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amzallag E, Panchadsaram T, Girard M, Lecluyse V, Couture E, D'Aragon F, Kandelman S, Turgeon AF, Jodoin C, Beaulieu P, Richebe P, Carrier FM. Pulmonary complications and mortality among COVID-19 patients undergoing a surgery: a multicentre cohort study. BMJ Open. 2024 Nov 21;14(11):e090158. doi: 10.1136/bmjopen-2024-090158. PMID 39578040
- [Derived] Carrier FM, Amzallag E, Lecluyse V, Cote G, Couture EJ, D'Aragon F, Kandelman S, Turgeon AF, Deschamps A, Nitulescu R, Djade CD, Girard M, Beaulieu P, Richebe P. Postoperative outcomes in surgical COVID-19 patients: a multicenter cohort study. BMC Anesthesiol. 2021 Jan 12;21(1):15. doi: 10.1186/s12871-021-01233-9. PMID 33435887